CLINICAL TRIAL: NCT06787482
Title: Open Label, Interventional Single Arm Study Evaluating a New Peptide Therapy for Retinal Diseases: AMD, Diabetic Retinopathy, and Dystrophies
Brief Title: Evaluating a New Peptide Therapy for Retinal Diseases: AMD, Diabetic Retinopathy, and Dystrophies
Acronym: Retino
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ace Cells Lab Limited (Industry)
Collaborators: European Wellness Academy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE_Retino_EG
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Retinitis Pigmentosa (RP); Age Related Macular Degeneration; Diabetic Retinopathy
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: The study should enroll 25 participants, rounded to 30 participants to ensure adequate power after accounting for variability and potential dropouts
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- administer 1 ml of Ace Retino 4 times daily for 6 months,safety evaluation (Active Comparator): Primary Objective: Evaluate the safety and tolerability of ACE Retino in individuals with RP.
  Interventions: Dietary Supplement: ACE Retino
- test efficacy for ACE Retino 1 ml 4times daily sublingual for 6 months (Experimental): Assess the efficacy of ACE Retino in improving retinal structure and function. Explore the potential for photoreceptor and retinal pigment epithelial (RPE) regeneration.
  Interventions: Dietary Supplement: ACE Retino

INTERVENTIONS:
Dietary Supplement: ACE Retino — 1 ml sublingually self administer / 4 times/day for 6 months

SUMMARY:
Summary of the Study This clinical trial evaluates a novel peptide-based therapy for treating retinal dystrophies, age-related macular degeneration (AMD), and diabetic retinopathy (DR). The therapy consists of peptides derived from fetal tissues, mesenchymal stem cells (MSCs), and bioactive growth factors, administered sublingually for systemic absorption.

Study Objectives:

Primary Objectives: Assess safety and tolerability, and evaluate the therapy's effects on retinal function and structure.

Secondary Objectives: Explore improvements in visual acuity, retinal thickness, vascular health, and disease biomarkers.

Study Design:

Type: Open-label, single-arm interventional study. Duration: 12 months.

Participants: 150 adults, divided into three cohorts:

Retinal dystrophies. AMD (dry and wet forms). DR (moderate NPDR and PDR).

Intervention:

A sublingual solution containing peptides and growth factors, taken 4 times daily.

Outcome Measures:

Primary Outcomes: Safety (adverse events) and tolerability (treatment adherence).

Secondary Outcomes:

Functional: Visual acuity and field sensitivity improvements. Structural: Retinal thickness and vascular health. Biomarkers: Serum VEGF, oxidative stress, and inflammatory markers.

Study Procedures:

Monthly follow-ups for safety monitoring, vision tests, retinal imaging (OCT, FA), and blood biomarker analysis.

Comprehensive evaluations at baseline, 6 months, and 12 months. Significance: The study aims to provide an innovative, non-invasive treatment for debilitating retinal conditions, potentially improving vision and retinal health through systemic therapy.

DETAILED DESCRIPTION:
Protocol for Evaluating a Novel Peptide-Based Therapy in Retinal Dystrophies, Age-Related Macular Degeneration, and Diabetic Retinopathy

Authors :

Mohamed Yasser Sayed Saif Prof of ophthalmology , Beni-Suef University Sherin Amer Family medicine consultant, Alaa Abdelkarim Endocrinology consultant , ACE Cells Lab Ahmed Tamer Sayed Saif Assistant Professor of ophthalmology, Fayoum University Passant Sayed Saif Assistant Professor of Ophthalmology, Misr University for Science and Technology

1. Background and Rationale Retinal diseases such as retinal dystrophies, age-related macular degeneration (AMD), and diabetic retinopathy (DR) are among the leading causes of blindness worldwide. These conditions result from different pathophysiological mechanisms but share common features like oxidative stress, chronic inflammation, and cellular degeneration.

   The novel therapy under evaluation consists of low molecular weight peptides derived from fetal tissues and mesenchymal stem cells (MSCs). The formulation also incorporates bioactive growth factors and essential peptides to support retinal health and regeneration. Sublingual administration ensures systemic absorption and avoids invasive delivery methods.
2. Objectives

<!-- -->

1. Primary Objectives

   * Assess the safety and tolerability of the peptide-based therapy.
   * Evaluate its effects on retinal function and structure in patients with retinal dystrophies, AMD, and DR.
2. Secondary Objectives

   * Explore improvements in visual function (acuity, field sensitivity).
   * Monitor changes in retinal thickness and vascular health.
   * Investigate its impact on disease biomarkers in the blood (e.g., VEGF, oxidative stress markers).
3. Study Design • Type: Open-label, interventional, single-arm study.

   * Duration: 12 months.
   * Participants: 150 participants, stratified equally into three cohorts:

     * Cohort 1: Retinal dystrophies (e.g., macular dystrophy, Stargardt disease).
     * Cohort 2: AMD (both dry and wet forms).
     * Cohort 3: Diabetic retinopathy (moderate NPDR and PDR).
4. Participants 4.1 Inclusion Criteria

   • Adults aged 18-80 years diagnosed with retinal dystrophies, AMD, or DR.

   • BCVA between 20/40 and 20/400 in the study eye.
   * Evidence of disease progression within the last 12 months (e.g., worsening visual acuity, OCT changes).
   * Stable systemic conditions allowing safe participation. 4.2 Exclusion Criteria
   * Active ocular infections or inflammation.
   * Recent ocular surgeries (within 3 months).
   * Co-existing advanced glaucoma or other retinal diseases.
   * Pregnancy or breastfeeding.
   * Hypersensitivity to components of the peptide formulation.
5. Intervention 5.1 Study Drug

   • Formulation: Sublingual solution containing peptides derived from fetal retinal, optic nerve, and neural tissues, MSC-derived peptides, and platelet growth factors.

   • Dosage: 1.0 mL sublingually, four times daily. 5.2 Administration

   • Self-administered by participants in the morning and evening.
6. Outcome Measures 6.1 Primary Outcomes • Safety:

   * Incidence and severity of adverse events (AEs) over 12 months. • Tolerability:
   * Adherence to treatment regimen and participant-reported discomfort. 6.2 Secondary Outcomes

<!-- -->

1. Functional Outcomes:

   o BCVA changes measured using ETDRS charts.
   * Visual field sensitivity improvement assessed by automated perimetry.
2. Structural Outcomes:

   o Retinal thickness and photoreceptor integrity evaluated by SD-OCT.

   o Vascular leakage and neovascularization assessed using fluorescein angiography (FA) and OCT angiography (OCTA).
3. Biochemical and Biomarker Outcomes:

   * Serum VEGF levels and oxidative stress markers.
   * Inflammatory cytokine profiles (e.g., IL-6, TNF-α).

7. Study Procedures 7.1 Screening Visit

1. Informed Consent: Participants will provide written consent after a detailed explanation of the study.

2. Baseline Assessments:

* Comprehensive medical and ocular history.
* BCVA measurement using ETDRS charts.
* SD-OCT imaging of retinal structure.
* FA and OCTA for vascular assessment.
* Blood sampling for biomarkers (VEGF, inflammatory cytokines). 7.2 Monthly Follow-Up Visits 1. Safety Monitoring: Documentation of AEs and systemic health assessment. 2. Ocular Assessments:
* BCVA measurement.
* SD-OCT imaging to monitor retinal thickness and integrity.
* OCTA and FA for vascular changes (if indicated). 7.3 Midpoint Visit (6 Months) 1. Repeat all baseline assessments, including biomarkers and electrophysiology (full-field ERG).

7.4 End-of-Study Visit (12 Months)

1. Comprehensive evaluation of functional, structural, and biochemical outcomes.
2. Participant feedback on therapy tolerability and perceived benefits.

8. Statistical Analysis

1. Sample Size Justification:

o Effect size and variability for BCVA improvement and retinal thickness changes are estimated from previous studies. A sample size of 150 ensures 80% power to detect a clinically meaningful difference at a 5% significance level.

2. Data Analysis Plan:

* Continuous variables (e.g., BCVA, OCT metrics) analyzed using paired t-tests or ANOVA.
* Proportions of responders (e.g., those with BCVA improvement ≥5 letters) analyzed using chi-square tests.
* Correlation analysis between biomarkers and functional outcomes.

  9. Ethical Considerations
  1. Regulatory Compliance:
* Conducted per the Declaration of Helsinki and ICH-GCP guidelines. 2. IRB Approval: Secured before study commencement. 3. Informed Consent: Participants provided detailed study information and signed consent forms.

  4. Data Confidentiality: All participant data anonymized and securely stored.

  10. References
  1. Wong WL, Su X, Li X, et al. Global prevalence of age-related macular degeneration and disease burden projection. Lancet Glob Health. 2014;2

     . doi:10.1016/S2214-109X(13)70145-1.
  2. Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010;376:124-36. doi:10.1016/S0140-6736(09)62124-3.
  3. Scholl HP, Strauss RW, Singh MS, et al. Emerging therapies for inherited retinal degeneration. Sci Transl Med. 2016;8:368rv6. doi:10.1126/scitranslmed.aaf2838.
  4. Ciulla TA, Amador AG, Zinman B. Diabetic retinopathy and diabetic macular edema: pathophysiology, screening, and novel therapies. Diabetes Care. 2003;26(9):2653-64. doi:10.2337/diacare.26.9.2653.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-65 years with a confirmed genetic or clinical diagnosis of RP.

  * Visual acuity of ≥1/60 in at least one eye.
  * Stable ocular and systemic condition over the past six months.
  * Ability to provide written informed consent

Exclusion Criteria:

* • Significant ocular comorbidities (e.g., advanced glaucoma, diabetic retinopathy).

  * Recent ocular surgery (within six months) or current use of investigational drugs.
  * Systemic conditions affecting study outcomes (e.g., uncontrolled diabetes, autoimmune diseases).
  * Pregnancy or lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in BVCA | 3 months
  change in BCVA (best-corrected visual acuity). The calculation is based on detecting a clinically meaningful improvement in BCVA using a paired design (before and after treatment within the same subjects).

SECONDARY OUTCOMES:
change in OCT | 3 months
  change in OCT curves and numbers based on before and after results

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Passant Sayed Saif, PhD ophthalmology, Principal Investigator — Associate prof of Ophthalmology Misr University for science and technology; Dr. Mohammed Yasser Sayed Saif, PhD Ophthalmology, Principal Investigator — Dean of NILES Prof of Ophthalmology Beni-Suef University; Dr. Alaa Abdelkarim Mohammed, MRCPUK Endocirnology, Principal Investigator — ACE Cells Lab Limited Chief Medical Consultant; Dr. Ahmed Tamer Sayed Saif, PhD Ophthalmology, Principal Investigator — Chairman of Ophthalmology department Associate prof of Ophthalmology Fayoum university; DR. Mike Chan, stem cells expert, Study Chair — European Wellness Academy
Locations (2):
- Egypt (2):
  - Dr. Seif Clinic, Cairo
  - British Center for Regeerative medicne (Cairo), Giza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.ace-cells.co.uk